CLINICAL TRIAL: NCT00089713
Title: Effect of ALT-711 in Combination With Fixed-Dose Hydrochlorothiazide Therapy on Systolic Blood Pressure in Hypertensive Patients
Brief Title: Systolic Pressure Efficacy and Safety Trial of Alagebrium (SPECTRA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-711-0320
Record Dates: First submitted 2004-08-10; First posted 2004-08-12 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2005-06

CONDITIONS: Hypertension
Keywords: antihypertensive agents/therapeutic use; hypertension/drug therapy; blood pressure
MeSH Terms: conditions — Hypertension | interventions — alagebrium

INTERVENTIONS:
Drug: alagebrium chloride (ALT-711)

SUMMARY:
This study comprises a 3- to 6-week hydrochlorothiazide run in phase, followed by a 12 week double-blind treatment phase, followed by a 2 week single-blind follow-up hydrochlorothiazide treatment phase. The combined total duration of patient participation is approximately 17-20 weeks. Four double-blind treatment groups approximately equal in size (98) will comprise the study population: placebo or various alagebrium dose groups (10, 50, or 150 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 45 years of age with uncontrolled systolic hypertension measured by office cuff and by an ambulatory blood pressure monitoring device
* Willingness to be taken off any current antihypertensive treatment to be placed on hydrochlorothiazide in combination with study medication.

Exclusion Criteria:

* Any significant history, systemic illnesses, or medical condition(s) that could lead to difficulty complying with the protocol or that could confound interpretation of the data.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Milan Kovacevic, MD, PhD, Study Director — Synvista Therapeutics, Inc
Locations (1):
- Alteon Inc., Parsippany, New Jersey, United States

REFERENCES:
- [Background] Kass DA, Shapiro EP, Kawaguchi M, Capriotti AR, Scuteri A, deGroof RC, Lakatta EG. Improved arterial compliance by a novel advanced glycation end-product crosslink breaker. Circulation. 2001 Sep 25;104(13):1464-70. doi: 10.1161/hc3801.097806. PMID 11571237
- [Background] Asif M, Egan J, Vasan S, Jyothirmayi GN, Masurekar MR, Lopez S, Williams C, Torres RL, Wagle D, Ulrich P, Cerami A, Brines M, Regan TJ. An advanced glycation endproduct cross-link breaker can reverse age-related increases in myocardial stiffness. Proc Natl Acad Sci U S A. 2000 Mar 14;97(6):2809-13. doi: 10.1073/pnas.040558497. PMID 10706607
- [Background] Wolffenbuttel BH, Boulanger CM, Crijns FR, Huijberts MS, Poitevin P, Swennen GN, Vasan S, Egan JJ, Ulrich P, Cerami A, Levy BI. Breakers of advanced glycation end products restore large artery properties in experimental diabetes. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4630-4. doi: 10.1073/pnas.95.8.4630. PMID 9539789
- [Background] Vaitkevicius PV, Lane M, Spurgeon H, Ingram DK, Roth GS, Egan JJ, Vasan S, Wagle DR, Ulrich P, Brines M, Wuerth JP, Cerami A, Lakatta EG. A cross-link breaker has sustained effects on arterial and ventricular properties in older rhesus monkeys. Proc Natl Acad Sci U S A. 2001 Jan 30;98(3):1171-5. doi: 10.1073/pnas.98.3.1171. PMID 11158613
- [Background] Chobanian AV. Control of hypertension--an important national priority. N Engl J Med. 2001 Aug 16;345(7):534-5. doi: 10.1056/NEJM200108163450709. No abstract available. PMID 11519509
- [Background] Hyman DJ, Pavlik VN. Characteristics of patients with uncontrolled hypertension in the United States. N Engl J Med. 2001 Aug 16;345(7):479-86. doi: 10.1056/NEJMoa010273. PMID 11519501
- [Background] Wilkinson IB, Webb Christison DJ, Cockcroft JR. Isolated systolic hypertension: a radical rethink. It's a risk factor that needs treatment, especially in the over 50s. BMJ. 2000 Jun 24;320(7251):1685. doi: 10.1136/bmj.320.7251.1685. No abstract available. PMID 10864525
- [Background] Brownlee M, Vlassara H, Kooney A, Ulrich P, Cerami A. Aminoguanidine prevents diabetes-induced arterial wall protein cross-linking. Science. 1986 Jun 27;232(4758):1629-32. doi: 10.1126/science.3487117.
- [Background] Neaton JD, Wentworth D. Serum cholesterol, blood pressure, cigarette smoking, and death from coronary heart disease. Overall findings and differences by age for 316,099 white men. Multiple Risk Factor Intervention Trial Research Group. Arch Intern Med. 1992 Jan;152(1):56-64. PMID 1728930
- [Background] Liu J, Masurekar MR, Vatner DE, Jyothirmayi GN, Regan TJ, Vatner SF, Meggs LG, Malhotra A. Glycation end-product cross-link breaker reduces collagen and improves cardiac function in aging diabetic heart. Am J Physiol Heart Circ Physiol. 2003 Dec;285(6):H2587-91. doi: 10.1152/ajpheart.00516.2003. Epub 2003 Aug 28. PMID 12946933